CLINICAL TRIAL: NCT01498237
Title: A Pilot Study of Photoacoustic Endoscopy in Endometrial Cancer
Brief Title: Photoacoustic Endoscopy in Endometrial Cancer
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Need to obtain IDE prior to commencement of study
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201102405
Record Dates: First submitted 2011-12-12; First posted 2011-12-23 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Endometrial Cancer; Benign Neoplasm of Body of Uterus
Keywords: Photoacoustic endoscopy
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Photoacoustic endoscopy (Experimental): This is a one-arm, feasibility study to determine how well the experimental procedure photoacoustic endoscopy will evaluate the human endometrial cavity in vivo.
  Interventions: Device: Photoacoustic endoprobe; Procedure: Photoacoustic endoscopy

INTERVENTIONS:
Device: Photoacoustic endoprobe — The PAE assessment will be performed in the operating room following strict sterile technique. PAE is performed immediately prior to the planned surgery. Participants are prepped following standard protocol. Length of the endometrial cavity is determined by a uterine sound. Endocervix is dilated as needed to allow passage of the PAE probe. The PAE probe will be advanced to the uterine fundus. Images will be obtained during withdrawal of the PAE probe from fundus to the os. Recorded images will allow computer assisted image analysis and functional measurements to be performed. Duration and difficulty of the procedure will be recorded. Comments and complications will be specifically noted.
  Other Names: There are no other interventions.
Procedure: Photoacoustic endoscopy — Photoacoustic endoscopy probe will be inserted into the endometrial canal to the uterine fundus and images will be obtained during the withdrawal of the probe from the fundus to the endocervical os.
  Other Names: There are no other interventions.

SUMMARY:
The purpose of this research study is to evaluate whether a new technology called intrauterine photoacoustic endoscopy (PAE) can be used to evaluate the inner lining of the uterus.

DETAILED DESCRIPTION:
The investigators will evaluate whether this technology can be used and also try to obtain photoacoustic images and functional data (oxygen contents, blood vessel characteristics, etc) of the uterine lining to assess its appearance in women with and without cancer of the endometrium. Currently, it is difficult for physicians to know whether or not tumors of the endometrium have invaded and spread to other organs without performing an extended surgery called a staging operation (removal of the lymph nodes or glands that drain the uterus to assess under the microscope whether or not the cancer has spread). Our long term goal is to use this new photoacoustic (PA) technology to improve detection of occult metastatic disease. Occult disease is defined as tumor which cannot be seen without the use of imaging techniques. and possibly avoid the need of extended operations. All of this could result in better care for patients with endometrial cancer and other gynecologic problems.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with benign gynecologic pathology (N=10) or biopsy proven endometrial cancer (N=10) who will undergo hysterectomy.
* Participants must be ≥ 18 years of age.
* Subjects of reproductive potential must have a negative pregnancy test prior to study photoacoustic endoscopy procedure and hysterectomy.
* Subjects must be able understand and willing to sign a written informed consent form.

Exclusion Criteria:

* Subjects with contraindications for general anesthesia or hysterectomy.
* Subjects with evidence of active pelvic inflammatory disease or purulent cervicitis.
* Subjects with prior endometrial ablation procedures.
* Gross tumoral involvement of the cervix or lower genital tract precluding cervical dilatation and endometrial sounding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of using the device to image endometrial cancer | 12 months or less
  Feasibility of using this novel device to image endometrial cancer is our primary objective. The frequency of success in obtaining images, overall and per group, will be presented and binomial success rates with 95% confidence interval estimates will be calculated. Besides the overall success rates, graphical and tabular summaries of the feasibility across patient demographic and clinical characteristics will be created.

CONTACTS AND LOCATIONS:
Overall Officials: Israel Zighelboim, MD, Principal Investigator — Washington University School of Medicine

REFERENCES:
- [Background] Morrow CP, Bundy BN, Kurman RJ, Creasman WT, Heller P, Homesley HD, Graham JE. Relationship between surgical-pathological risk factors and outcome in clinical stage I and II carcinoma of the endometrium: a Gynecologic Oncology Group study. Gynecol Oncol. 1991 Jan;40(1):55-65. doi: 10.1016/0090-8258(91)90086-k. PMID 1989916
- [Background] Kilgore LC, Partridge EE, Alvarez RD, Austin JM, Shingleton HM, Noojin F 3rd, Conner W. Adenocarcinoma of the endometrium: survival comparisons of patients with and without pelvic node sampling. Gynecol Oncol. 1995 Jan;56(1):29-33. doi: 10.1006/gyno.1995.1005. PMID 7821843
- [Background] Cragun JM, Havrilesky LJ, Calingaert B, Synan I, Secord AA, Soper JT, Clarke-Pearson DL, Berchuck A. Retrospective analysis of selective lymphadenectomy in apparent early-stage endometrial cancer. J Clin Oncol. 2005 Jun 1;23(16):3668-75. doi: 10.1200/JCO.2005.04.144. Epub 2005 Feb 28. PMID 15738538
- [Background] Chan JK, Cheung MK, Huh WK, Osann K, Husain A, Teng NN, Kapp DS. Therapeutic role of lymph node resection in endometrioid corpus cancer: a study of 12,333 patients. Cancer. 2006 Oct 15;107(8):1823-30. doi: 10.1002/cncr.22185. PMID 16977653
- [Background] Keys HM, Roberts JA, Brunetto VL, Zaino RJ, Spirtos NM, Bloss JD, Pearlman A, Maiman MA, Bell JG; Gynecologic Oncology Group. A phase III trial of surgery with or without adjunctive external pelvic radiation therapy in intermediate risk endometrial adenocarcinoma: a Gynecologic Oncology Group study. Gynecol Oncol. 2004 Mar;92(3):744-51. doi: 10.1016/j.ygyno.2003.11.048. PMID 14984936
- [Background] Jemal A, Siegel R, Ward E, Hao Y, Xu J, Thun MJ. Cancer statistics, 2009. CA Cancer J Clin. 2009 Jul-Aug;59(4):225-49. doi: 10.3322/caac.20006. Epub 2009 May 27. PMID 19474385
- [Background] ASTEC study group; Kitchener H, Swart AM, Qian Q, Amos C, Parmar MK. Efficacy of systematic pelvic lymphadenectomy in endometrial cancer (MRC ASTEC trial): a randomised study. Lancet. 2009 Jan 10;373(9658):125-36. doi: 10.1016/S0140-6736(08)61766-3. Epub 2008 Dec 16. PMID 19070889
- [Background] Benedetti Panici P, Basile S, Maneschi F, Alberto Lissoni A, Signorelli M, Scambia G, Angioli R, Tateo S, Mangili G, Katsaros D, Garozzo G, Campagnutta E, Donadello N, Greggi S, Melpignano M, Raspagliesi F, Ragni N, Cormio G, Grassi R, Franchi M, Giannarelli D, Fossati R, Torri V, Amoroso M, Croce C, Mangioni C. Systematic pelvic lymphadenectomy vs. no lymphadenectomy in early-stage endometrial carcinoma: randomized clinical trial. J Natl Cancer Inst. 2008 Dec 3;100(23):1707-16. doi: 10.1093/jnci/djn397. Epub 2008 Nov 25. PMID 19033573
- [Background] ASTEC/EN.5 Study Group; Blake P, Swart AM, Orton J, Kitchener H, Whelan T, Lukka H, Eisenhauer E, Bacon M, Tu D, Parmar MK, Amos C, Murray C, Qian W. Adjuvant external beam radiotherapy in the treatment of endometrial cancer (MRC ASTEC and NCIC CTG EN.5 randomised trials): pooled trial results, systematic review, and meta-analysis. Lancet. 2009 Jan 10;373(9658):137-46. doi: 10.1016/S0140-6736(08)61767-5. Epub 2008 Dec 16. PMID 19070891
- [Background] Creasman W. Revised FIGO staging for carcinoma of the endometrium. Int J Gynaecol Obstet. 2009 May;105(2):109. doi: 10.1016/j.ijgo.2009.02.010. Epub 2009 Apr 3. No abstract available. PMID 19345353
- [Background] Zerbe MJ, Bristow R, Grumbine FC, Montz FJ. Inability of preoperative computed tomography scans to accurately predict the extent of myometrial invasion and extracorporal spread in endometrial cancer. Gynecol Oncol. 2000 Jul;78(1):67-70. doi: 10.1006/gyno.2000.5820. PMID 10873413
- [Background] Connor JP, Andrews JI, Anderson B, Buller RE. Computed tomography in endometrial carcinoma. Obstet Gynecol. 2000 May;95(5):692-6. doi: 10.1016/s0029-7844(99)00626-2. PMID 10775731
- [Background] Hricak H, Rubinstein LV, Gherman GM, Karstaedt N. MR imaging evaluation of endometrial carcinoma: results of an NCI cooperative study. Radiology. 1991 Jun;179(3):829-32. doi: 10.1148/radiology.179.3.2028000.
- [Background] Cabrita S, Rodrigues H, Abreu R, Martins M, Teixeira L, Marques C, Mota F, de Oliveira CF. Magnetic resonance imaging in the preoperative staging of endometrial carcinoma. Eur J Gynaecol Oncol. 2008;29(2):135-7. PMID 18459546
- [Background] Horowitz NS, Dehdashti F, Herzog TJ, Rader JS, Powell MA, Gibb RK, Grigsby PW, Siegel BA, Mutch DG. Prospective evaluation of FDG-PET for detecting pelvic and para-aortic lymph node metastasis in uterine corpus cancer. Gynecol Oncol. 2004 Dec;95(3):546-51. doi: 10.1016/j.ygyno.2004.08.009. PMID 15581961
- [Background] Park JY, Kim EN, Kim DY, Suh DS, Kim JH, Kim YM, Kim YT, Nam JH. Comparison of the validity of magnetic resonance imaging and positron emission tomography/computed tomography in the preoperative evaluation of patients with uterine corpus cancer. Gynecol Oncol. 2008 Mar;108(3):486-92. doi: 10.1016/j.ygyno.2007.11.044. Epub 2008 Jan 16. PMID 18201753
- [Background] Zhang HF, Maslov K, Stoica G, Wang LV. Functional photoacoustic microscopy for high-resolution and noninvasive in vivo imaging. Nat Biotechnol. 2006 Jul;24(7):848-51. doi: 10.1038/nbt1220. Epub 2006 Jun 25. PMID 16823374
- [Background] Wang X, Pang Y, Ku G, Xie X, Stoica G, Wang LV. Noninvasive laser-induced photoacoustic tomography for structural and functional in vivo imaging of the brain. Nat Biotechnol. 2003 Jul;21(7):803-6. doi: 10.1038/nbt839. Epub 2003 Jun 15. PMID 12808463
- [Background] Wang LV. Prospects of photoacoustic tomography. Med Phys. 2008 Dec;35(12):5758-67. doi: 10.1118/1.3013698. PMID 19175133
- [Background] Yang JM, Maslov K, Yang HC, Zhou Q, Shung KK, Wang LV. Photoacoustic endoscopy. Opt Lett. 2009 May 15;34(10):1591-3. doi: 10.1364/ol.34.001591. PMID 19448831
- [Background] Wang LV. Multiscale photoacoustic microscopy and computed tomography. Nat Photonics. 2009 Aug 29;3(9):503-509. doi: 10.1038/nphoton.2009.157. PMID 20161535
- [Background] Ku G, Maslov K, Li L, Wang LV. Photoacoustic microscopy with 2-microm transverse resolution. J Biomed Opt. 2010 Mar-Apr;15(2):021302. doi: 10.1117/1.3339912. PMID 20459224
- [Background] Maslov K, Zhang HF, Hu S, Wang LV. Optical-resolution photoacoustic microscopy for in vivo imaging of single capillaries. Opt Lett. 2008 May 1;33(9):929-31. doi: 10.1364/ol.33.000929. PMID 18451942
- [Background] Song KH, Kim C, Cobley CM, Xia Y, Wang LV. Near-infrared gold nanocages as a new class of tracers for photoacoustic sentinel lymph node mapping on a rat model. Nano Lett. 2009 Jan;9(1):183-8. doi: 10.1021/nl802746w. PMID 19072058
- [Background] Chang KJ, Nguyen P, Erickson RA, Durbin TE, Katz KD. The clinical utility of endoscopic ultrasound-guided fine-needle aspiration in the diagnosis and staging of pancreatic carcinoma. Gastrointest Endosc. 1997 May;45(5):387-93. doi: 10.1016/s0016-5107(97)70149-4. PMID 9165320
- [Background] Menzel J, Domschke W. Gastrointestinal miniprobe sonography: the current status. Am J Gastroenterol. 2000 Mar;95(3):605-16. doi: 10.1111/j.1572-0241.2000.01832.x. PMID 10710047
- [Background] Tearney GJ, Brezinski ME, Bouma BE, Boppart SA, Pitris C, Southern JF, Fujimoto JG. In vivo endoscopic optical biopsy with optical coherence tomography. Science. 1997 Jun 27;276(5321):2037-9. doi: 10.1126/science.276.5321.2037. PMID 9197265
- [Background] Yun SH, Tearney GJ, Vakoc BJ, Shishkov M, Oh WY, Desjardins AE, Suter MJ, Chan RC, Evans JA, Jang IK, Nishioka NS, de Boer JF, Bouma BE. Comprehensive volumetric optical microscopy in vivo. Nat Med. 2006 Dec;12(12):1429-33. doi: 10.1038/nm1450. Epub 2006 Nov 19. PMID 17115049
- [Background] Kiesslich R, Burg J, Vieth M, Gnaendiger J, Enders M, Delaney P, Polglase A, McLaren W, Janell D, Thomas S, Nafe B, Galle PR, Neurath MF. Confocal laser endoscopy for diagnosing intraepithelial neoplasias and colorectal cancer in vivo. Gastroenterology. 2004 Sep;127(3):706-13. doi: 10.1053/j.gastro.2004.06.050. PMID 15362025
- [Background] Hu S, Wang LV. Photoacoustic imaging and characterization of the microvasculature. J Biomed Opt. 2010 Jan-Feb;15(1):011101. doi: 10.1117/1.3281673. PMID 20210427
- [Background] Piantadosi S. Translational clinical trials: an entropy-based approach to sample size. Clin Trials. 2005;2(2):182-92. doi: 10.1191/1740774505cn078oa. PMID 16279140
- [Background] American National Standards Institute. Laser Institute of America.American National Standards for Safe Use of Lasers ANSI Z136.1 - 2007. American National Standards Institute, Inc. New York NY, 2007
- See also: Alvin J.Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu